CLINICAL TRIAL: NCT05395364
Title: A Health Promotion Intervention for Vulnerable School - Children and Families: a Cluster-randomized Trial
Brief Title: A Health Promotion Intervention for Vulnerable School
Acronym: BeE-school
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minho (Other)
Responsible Party: Principal Investigator, Helena Rafaela Vieira do Rosario, Principal Investigator, PhD, University of Minho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UMinho
Record Dates: First submitted 2022-05-16; First posted 2022-05-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Health Promotion; Noncommunicable Diseases; Child Development; Life Style
MeSH Terms: conditions — Obesity; Noncommunicable Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No intervention will occur.
- Intervention (Experimental): An intervention program based on the promotion of health literacy and lifestyles, specifically on children's: 1-health literacy and infodemic resilience; 2- lifestyles (e.g. dietary intake, 24h-movement behaviour); 3-overweight and obesity; 4-blood pressure.
  Interventions: Behavioral: Intervention program BeE-school

INTERVENTIONS:
Behavioral: Intervention program BeE-school — The intervention program will be co-developed and directed to school professionals. It will be based on the promotion of health literacy and lifestyles.
  Arms: Intervention

SUMMARY:
The BeE-school (Be Empowered in school) is a cluster-randomised trial that addresses the complexity of the social challenge (vulnerable school-age children). It aims to analyse the effectiveness of the intervention program, based on the promotion of health literacy and lifestyles, specifically on children's: 1-health literacy and infodemic resilience (Aim 1); 2- lifestyles (e.g. dietary intake, 24hmovement behaviour) (Aim 2); 3-overweight and obesity (Aim 3); 4-blood pressure (Aim 4). The project converges multiple disciplines (e.g. public health, informatics, law) and researchers with proven expertise in these fields to provide comprehensive and innovative answers. 478 children (6 schools) aged 6-12years old will participate in this cluster-randomised trial, having schools as the unit of randomisation, assigned into intervention (239-3schools) and the control arm (239 - 3 schools). This project will perform a social listening (online and offline) and bottom-up approach to tackling NCDs, focusing on health literacy and health promotion and recognising children's systems in daily life (e.g. family, teachers). Stakeholders' involvement goes far beyond a merely consultative approach; the researchers are committed to a genuine codevelopment process. Data collection includes sociodemographics, health literacy and infodemic resilience, dietary intake and children's 24-h movement behaviour (e.g. accelerometry), anthropometry (e.g. weight, height and waist circumference) and blood pressure. Data collection will occur at baseline and after the intervention (follow-up, 6 months after the beginning of the intervention). Expected outputs and outcomes include the creation of a model for characterising NCDs and health topics based on artificial intelligence techniques (e.g. deep learning, and social network analysis methods); improved health literacy and infodemic resilience of children, families and teachers; enhanced children's lifestyles (e.g. dietary intake, 24-h movement behaviour); reduction of NCDs' physical risk factors (e.g. overweight, raised blood pressure); feasible intervention program about health promotion and NCDs' prevention for school-aged children with vulnerabilities, and advocacy- policies about health promotion and NCDs' prevention.

ELIGIBILITY:
Inclusion Criteria:

* Children from TEIP schools
* Ages between 5 to 12 years old

Exclusion Criteria:

* Children/families who don't speak/understand Portuguese

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 735 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Overweight and obesity | 6 months
  Anthropometry (weight and height will be combined to report BMI in kg/m^2)
Risk of high blood pressure | 6 months
  Blood pressure monitoring (systolic and diastolic blood pressure)
Health literacy | 6 months
  European health literacy questionnaire (HLS19-Q12-PT) - range between 0 and 100. The cut-offs for categorizing health literacy were based on the following positions: below 50; between 50 and 66.66; between 66.67 and 83.33; above 83.34. These cut-offs allowed the definition of the same categories as in the HLS-EU study: "inadequate" and "problematic" (low health literacy), "adequate" and "excellent" (high health literacy).
Dietary intake | 6 months
  Dietary intake (24h dietary recall) - recall the intake of foods in the previous day.
Physical activity | 6 months
  Physical activity will be assessed using Actigraph GT3X+ accelerometers (ActiGraph, Pensacola, Florida, USA) over a usual week (24 h/day over 7 days - except for water activities). These devices are small, light and unobtrusive, worn on the wrist, and their validity and utility have previously been established in children. For this study, one count per minute will be converted into light, moderate or vigorous activity. Parents will be asked to fill in an activity monitor log with the times that the accelerometers were removed and put back onto the child.
Sedentary behavior | 6 months
  Sedentary behavior will be assessed using Actigraph GT3X+ accelerometers (ActiGraph, Pensacola, Florida, USA) over a usual week (24 h/day over 7 days - except for water activities). These devices are small, light and unobtrusive, worn on a belt around the waist, and their validity and utility have previously been established in children. For this study values below 100 counts/min will be considered as sedentary behaviour. Parents will be asked to fill in an activity monitor log with the times that the accelerometers were removed and put back onto the child.
Sleep time | 6 months
  Sleep time will be assessed using Actigraph GT3X+ accelerometers (ActiGraph, Pensacola, Florida, USA) over a usual week (24 h/day over 7 days - except for water activities). These devices are small, light and unobtrusive, worn on a belt around the waist, and their validity and utility have previously been established in children. Parents will be asked to fill in an activity monitor log with the times that the accelerometers were removed and put back onto the child.
Sleep quality | 6 months
  Sleep quality will be assessed with the Portuguese Children's Sleep Habits Questionnaire, which along with Actigraph seems to better inform clinical practice and research on a child's sleep. The Children's Sleep Habits Questionnaire has the following dimensions: bedtime behavior and sleep onset; sleep duration; anxiety around sleep; behavior occurring during sleep and night wakings; sleep-disordered breathing; parasomnias; and morning waking/daytime sleepiness. Parents are asked to recall sleep behaviors occurring over a "typical" recent week. Items are rated on a three-point scale: "usually" if the sleep behavior occurred five to seven times/week; "sometimes" for two to four times/week; and "rarely" for zero to one time/week.

CONTACTS AND LOCATIONS:
Overall Officials: Rafaela D Rosário, PhD, Principal Investigator — University of Minho
Locations (1):
- Ana Duarte, Braga, Portugal

IPD SHARING:
Plan to Share IPD: No